CLINICAL TRIAL: NCT06862921
Title: Effects of Dıfferent Tournıques and Posıtıons on Paın, Anxıety Levels and Applıcatıon Success in Perıpheral Intravenous Catheter Applıcatıon: a Randomızed Controlled Study
Acronym: CATHETER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Şerife Kelle Dikbaş, MSC, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: Uskudar University; Clinical Research Ethics Commi (Registry Identifier: 2024/74)
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Tourniquets; INTRAVENOUS CATHETER APPLICATION
Keywords: Peripheral Catheterization; tourniquet; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Group 1 (Experimental): standard tourniquet in the supine position
  Interventions: Other: Control
- Experimental Group 2 (Experimental): sphygmomanometer at 60 mmHg pressure in the fawler position
  Interventions: Other: Control
- Experimental Group 3 (Experimental): sphygmomanometer at 60 mmHg pressure in the supine position
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — fawler position using a standard tourniquet

SUMMARY:
Aim:

The aim of this study was to investigate the effect of different tourniquet and position on pain, anxiety level and success of peripheral intravenous catheter (PIC) application.

Design:

Randomized controlled experimental design.

DETAILED DESCRIPTION:
Aim:

The aim of this study was to investigate the effect of different tourniquet and position on pain, anxiety level and success of peripheral intravenous catheter (PIC) application.

Primary purpose:investigate the effect of different tourniquet and position on pain, Secondary purpose:investigate the effect of different tourniquet and position on anxiety level and success of peripheral intravenous catheter (PIC) application.

Design:

Randomized controlled experimental design.

Methods:

The randomized controlled experimental design study was conducted with 110 adult patients in the orthopedic department of a Training and Research Hospital between May 2024 and July 2024. Data were collected using the Patient Information Form, Visual Infusion Phlebitis Diagnostic Scale, Infiltration Scale, Visual Pain Scale, and Facial Anxiety Scale. PIC was applied to patients in the "Experimental Group 1" using a standard tourniquet in the supine position, to patients in the "Experimental Group 2" using a sphygmomanometer at 60 mmHg pressure in the fawler position, and to patients in the "Experimental Group 3" using a sphygmomanometer at 60 mmHg pressure in the supine position. In the control group, a peripheral intravenous catheter was applied in the fawler position using a standard tourniquet. Patients were asked to evaluate the level of pain and anxiety before and after the application. The patients were followed up for phlebitis and extravasation findings at eight-hour intervals after the application. Except for complications requiring removal of the peripheral intravenous catheter during follow-up, the PIC was removed 96 hours after application. The results were evaluated at 95% confidence intervals with a significance level of p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patient

  1. Volunteering to participate in the research
  2. Be between the ages of 18-64,
  3. The planned length of hospitalization is not less than 96 hours.

     Exclusion Criteria:

     In the patient

  <!-- -->

  1. Coagulation, hematologic and hydration problems
  2. Oncological, allergic diseases, any incision or scar tissue in the antecubital area, presence of complications due to a previously opened catheter, presence of pain, hematoma, ecchymosis in the application area, or presence of any other injection in the antecubital area on treatment days,
  3. The presence of an obstacle (such as mastectomy) in the arm to be treated.

     Expulsion criteria from the study:

  <!-- -->

  1. Dislodgement of the peripheral intravenous catheter for any reason.
  2. Failure of peripheral intravenous catheter placement more than twice.
  3. Discharge of the patient from the hospital.

Ages: 18 Weeks to 64 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Infusion Phlebitis Diagnostic Scale | 3 month
  This scale developed by Schultze and Gallant (2006) was published by the Infusion Nurses Society (2006) and is a widely used scale in the clinical evaluation of infusion phlebitis. Phlebitis assessment was evaluated by the investigator using the VIFFS once every eight hours until the PIC was removed and recorded on the patient follow-up form.
Infiltration Scale (IS) | 3 month
  Infiltration Scale (IS): This scale was published by the Intravenous Nurses Association (2006) and its psychometric properties were evaluated by Groll et al. Infiltration assessment was evaluated by the investigator using the IS once every eight hours until the PIC was removed and recorded on the patient follow-up form
Visual Pain Scale (VAS): | 3 month
  Visual Pain Scale (VAS): This scale was developed by Hayes and Patterson in 1921 and is used to assess pain intensity. Pain intensity is measured using a 10 cm visual scale; mean pain scores ranging from 0 to 10 are given. zero indicates the absence of pain, ten indicates the presence of severe pain. A VAS value of one to four indicates mild pain, five to six indicates moderate pain, and seven to ten indicates severe pain. The researcher asked the patient to indicate the severity of pain according to VAS before and after PIC placement and recorded the value on the patient follow-up form.
Facial Anxiety Scale (FAS) | 3 month
  Facial Anxiety Scale (FAS): The Turkish validity and reliability of the scale developed by McKinley, Coote, and Stein-Parbury (2003) was performed by İyigün, Pazar, and Taştan (2016). The Face Anxiety Scale is 11 × 42 cm in size. It consists of five different facial expressions, the leftmost facial expression indicates the absence of anxiety, while the level of anxiety increases from left to right. The FAS is scored from zero to five from left to right, respectively. A score of three on this scale indicates moderate anxiety, while a score of four and above indicates high anxiety. In this scale, the patient evaluates his/her own anxiety (McKinley 2004). The researcher showed the scale to the patient before and after PIC placement and asked the patient to evaluate which facial expression corresponded to his/her anxiety level and recorded the result on the patient follow-up form.Application of research

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Martyr Prof. Dr. İlhan Varank Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year

REFERENCES:
- [Background] Tran QK, Flanagan K, Fairchild M, Yardi I, Pourmand A. Nurses and Efficacy of Ultrasound-Guided Versus Traditional Venous Access: A Systemic Review and Meta-Analysis. J Emerg Nurs. 2022 Mar;48(2):145-158.e1. doi: 10.1016/j.jen.2021.12.003. Epub 2022 Feb 4. PMID 35125291
- [Background] Tran T, Lund SB, Nichols MD, Kummer T. Effect of two tourniquet techniques on peripheral intravenous cannulation success: A randomized controlled trial. Am J Emerg Med. 2019 Dec;37(12):2209-2214. doi: 10.1016/j.ajem.2019.03.034. Epub 2019 Mar 23. PMID 30948254